CLINICAL TRIAL: NCT00276575
Title: Phase I Study of Bevacizumab in Combination With Everolimus and Erlotinib in Advanced Cancer
Brief Title: Bevacizumab, Everolimus, and Erlotinib in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008048; DUMC-6026-05-6R1; GENENTECH-DUMC-6026-05-6R1; NOVARTIS-DUMC-6026-05-6R1; CDR0000449970 (Other: NCI)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Bevacizumab; Erlotinib Hydrochloride; Everolimus

ARMS (1):
- Bevacizumab, Everolimus, and Erlotinib (Experimental): Dose Level Dose Bevacizumab (mg/kg q2wks) Everolimus (mg daily) Erlotinib (mg daily) -1 5 5 ---
  1. 10 5 ---
  2. 10 10 ---
  3. 10* 10* 75
  4. 10* 10* 150
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Drug: everolimus

INTERVENTIONS:
Biological: bevacizumab
Drug: erlotinib hydrochloride
Drug: everolimus

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and everolimus may also block blood flow to the tumor. Giving everolimus and erlotinib together with bevacizumab may kill more tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of erlotinib and everolimus when given together with bevacizumab in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the maximum tolerated dose (MTD)/recommended phase II regimen of everolimus and erlotinib hydrochloride when given with bevacizumab in patients with advanced solid tumors.
* Evaluate safety of bevacizumab, everolimus, and erlotinib hydrochloride in these patients.

Secondary

* Describe the impact of this combination therapy on dermal wound angiogenesis and inhibition of vascular endothelial growth factor receptor 1 (VEGFR1), mTOR/p70S6K, and other related markers in granulation tissue.
* Evaluate clinical activity (partial response, complete response, or stable disease > 6 months) associated with this regimen.

OUTLINE: This is a dose-escalation study followed by a randomized study.

* Part 1: Patients receive bevacizumab IV on days 1 and 15 and oral everolimus and oral erlotinib hydrochloride* once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive escalating doses of everolimus or escalating doses of everolimus and erlotinib hydrochloride* until the maximum tolerated dose (MTD) is determined. Patients in part 2 of the study are treated at the MTD of everolimus and erlotinib hydrochloride.

NOTE: *The first cohort of patients receive bevacizumab and everolimus only until the MTD is determined, the subsequent cohorts of patients receive bevacizumab, everolimus, and erlotinib hydrochloride

* Part 2: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral everolimus once daily beginning on day 1, oral erlotinib hydrochloride once daily beginning on day 15, and bevacizumab IV once every 2 weeks beginning on day 15. Treatment continues in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive oral erlotinib hydrochloride once daily beginning on day 1, oral everolimus once daily beginning on day 15, and bevacizumab IV once every 2 weeks beginning on day 15. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy

  * Metastatic or unresectable disease
* Standard curative or palliative measures do not exist OR are no longer effective
* No CNS metastases
* No centrally-located non-small cell lung cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Leukocytes ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN (5 times ULN if known hepatic metastases)
* Urine protein to creatinine ratio ≤ 1.0 OR urine protein < 1 g by 24 hour urine collection
* Creatinine clearance ≥ 50 mL/min OR creatinine normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for up to 4 months after study treatment has stopped
* No uncontrolled hypertriglyceridemia (i.e., fasting serum triglyceride > 350 mg/dL)
* No uncontrolled hypercholesterolemia (i.e., fasting serum cholesterol > 300 mg/dL)
* No poorly controlled hypertension (i.e., blood pressure > 160/100 mm Hg)
* No poorly controlled or clinically significant atherosclerotic vascular disease
* No thrombosis within 6 months
* No venous thromboembolic event within 6 months
* No arterial thromboembolic events within 12 months
* No cerebrovascular accident or transient ischemic attack in past 12 months
* No myocardial infarction or unstable angina in past 12 months
* No clinically significant peripheral vascular disease in past 12 months
* No New York Heart Association class II-IV congestive heart failure

  * Atrial or supraventricular tachycardias well controlled with beta blocker or calcium channel blocker allowed
  * Chronic pacemaker use allowed
* No serious cardiac arrhythmia requiring medication
* No other clinically significant cardiovascular disease
* No hemoptysis > 1 tablespoon within 6 months
* No presence of bleeding diathesis
* No coagulopathy
* No presence of significant gastrointestinal (GI) disorders that would affect drug absorption
* No hemodynamically significant GI bleeding
* No history of intolerance to bevacizumab, everolimus, or erlotinib
* No other major bleeding event
* No ongoing or active infection
* No psychiatric illness or social situations that would limit safety or compliance with study requirements
* No other uncontrolled intercurrent illness

PRIOR CONCURRENT THERAPY:

* No angioplasty or cardiac or vascular stenting within the past 12 months
* No major surgery within past 28 days
* No other investigational agents within past 28 days
* No chemotherapy for cancer within past 21 days
* No biologic therapy for cancer within past 21 days
* No radiation therapy for cancer within past 21 days
* No hormonal therapy for cancer within past 21 days
* No minor surgical procedures within past 14 days
* No concurrent antiplatelet agents other than aspirin < 325 mg/day
* No use of statin drugs other than pravastatin or atorvastatin
* Initiation of blood pressure (BP) medication is permitted prior to study entry provided that BP < 150/90 mm Hg on 3 measurements over one week (study day -7 to 1) before starting treatment
* No concurrent grapefruit juice
* No concurrent therapeutic anticoagulation

  * Prophylactic low-dose anticoagulation for indwelling catheters is permitted
* No concurrent administration of any of the following drugs:

  * Nicardipine
  * Verapamil
  * Clotrimazole
  * Fluconazole
  * Itraconazole
  * Ketoconazole
  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Cisapride
  * Metoclopramide
  * Bromocriptine
  * Cimetidine
  * Danazol
  * HIV-protease inhibitors (e.g., ritonavir, indinavir)
  * Hypericum perforatum (St. John's wort)
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Diltiazem
  * Rifabutin
  * Rifapentine
  * Rifampin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-03; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Until study completion
  Its primary objective is to estimate the MTD/recommended phase II dose combination or regimen

SECONDARY OUTCOMES:
Safety | Until study completion
  endpoints will be evaluated in an exploratory fashion

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Bullock KE, Petros WP, Younis I, Uronis HE, Morse MA, Blobe GC, Zafar SY, Gockerman JP, Lager JJ, Truax R, Meadows KL, Howard LA, O'Neill MM, Broadwater G, Hurwitz HI, Bendell JC. A phase I study of bevacizumab (B) in combination with everolimus (E) and erlotinib (E) in advanced cancer (BEE). Cancer Chemother Pharmacol. 2011 Feb;67(2):465-74. doi: 10.1007/s00280-010-1507-6. Epub 2010 Nov 16. PMID 21079958